CLINICAL TRIAL: NCT04175483
Title: The Evaluation of Airway Dimension by Using Ultrasonography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201910015RINC
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2019-11

CONDITIONS: Subglottic Airway Diameter in Normal Adults

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: assessment of subglottic diameter by ultrasonography — assessment of subglottic diameter by ultrasonography

SUMMARY:
The aim of this study is to measure the dimension of airway in healthy Asian population. We recruit normal volunteer subjects aged more than 20 years old. Subglottic transverse diameter is measured and recorded by ultrasonography.

DETAILED DESCRIPTION:
The aim of this study is to measure the dimension of airway in healthy Asian population. We recruit normal volunteer subjects aged more than 20 years old. Subglottic transverse diameter is measured and recorded by ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy volunteers (aged more than 20 years) without pre-existing airway or respiratory diseases, neck tumors and a history of neck operation.

Exclusion Criteria:

* pre-existing airway or respiratory diseases, neck tumors and a history of neck operation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult healthy volunteers (aged more than 20 years) without pre-existing airway or respiratory diseases, neck tumors and a history of neck operation.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
transverse glottic diameter by ultrasonography | one day
  transverse glottic diameter by ultrasonography

CONTACTS AND LOCATIONS:
Locations (1):
- Wan-Ching Lien, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No